CLINICAL TRIAL: NCT06521983
Title: The Effect of Whole Body Vibration on Pain and Muscle Elasticity in Individuals With Hyperlordosis and Normal Lordosis
Brief Title: The Effect of Whole Body Vibration on Muscle Elasticity
Acronym: WBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Gönül Elpeze, Assistant Proffessor, Gaziantep Islam Science and Technology University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GİBTU-GE-VİBRATİON
Record Dates: First submitted 2024-07-10; First posted 2024-07-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Lordosis; Postural; Lordosis; Hyperlordosis
Keywords: Whole-body vibration; Lordosis; Hyperlordosis
MeSH Terms: conditions — Lordosis; Swayback

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LORDOSİS (Experimental): 30-40
  Interventions: Other: Whole body vibration
- HYPERLORDOSİS (Experimental): 40<
  Interventions: Other: Whole body vibration

INTERVENTIONS:
Other: Whole body vibration — Whole body vibration will be applied while standing with a frequency of 30 Hz and an intensity of 2 mm by vibration machine

SUMMARY:
This study examined the effect of whole-body vibration on pain and muscle elasticity in individuals with hyperlordosis and normal lordosis.

Flexible ruler for individuals' spinal curvatures (lumbar lordosis); back-lower back pain levels VAS; muscle elasticity Myoton Pro device; Physical functions will be evaluated with the Modified Oswestry low back pain scale.

DETAILED DESCRIPTION:
This study examined the effect of whole-body vibration on pain and muscle elasticity in individuals with hyperlordosis and normal lordosis.

Flexible ruler for individuals' spinal curvatures (lumbar lordosis); back-lower back pain levels VAS; muscle elasticity Myoton Pro device; Physical functions will be evaluated with the Modified Oswestry low back pain scale.

The viscoelasticity properties ( tone, stiffness, elasticity) of the Musculus Trapezius and Musculus Pectoralis were assessed with MyotonPro® (Myoton AS, Estonia) during prone position on both sides.

Individuals will be divided into two groups: hyperlordosis and normal lordosis. Whole body vibration will be applied twice a week for six weeks, with a frequency of 30 Hz and an intensity of 2 mm.

A total of 28 females and males (14 individuals for each group) with hyperlordosis (>40°) and normal lordosis participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Having pain >5 according to VAS measurement,
* Having normal lumbar lordosis angle between 30°-40°,
* Having hyperlordosis angle >40°

Exclusion Criteria:

* Having Scheurmann kyphosis, ,
* Having scoliosis (Cobb angle >10°),
* Having other congenital spine abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Muscle viscoelastic properties | 6 weeks
  muscle stiffness

SECONDARY OUTCOMES:
Pain level | 6 weeks
  Visual Analog Scale: between 0 -10 points; 0 (zero) no pain; 5 (five) Moderate pain; 10 (ten) Worst possible Pain

CONTACTS AND LOCATIONS:
Overall Officials: Gonul Elpeze, Principal Investigator — Gaziantep Islam Science and Technology University Physical Therapy and Rehabilitation Department
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No